CLINICAL TRIAL: NCT04024046
Title: Evaluation of the Impact of the Uqora Dietary Supplement Products on Urinary Tract Infection (UTI) Incidence in Women With Recurring UTIs
Brief Title: Uqora Supplements in Women With UTIs
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Hawthorne Effect Inc. (Other)
Collaborators: Uqora, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00034128
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control - Placebo: 1. Placebo Drink-Mix Daily for 180 days
  2. Placebo Capsules Daily for 180 days
  Interventions: Dietary Supplement: Uqora
- Group 1: 1. Uqora Drink-Mix Daily for 180 days
  2. Placebo Capsules Daily for 180 days
  Interventions: Dietary Supplement: Group1
- Group 2: 1. Uqora Drink-Mix Daily for 180 days
  2. Uqora Capsules Daily for 180 days
  Interventions: Dietary Supplement: Group 2

INTERVENTIONS:
Dietary Supplement: Uqora — Participants will receive 1 Placebo Drink-Mix and 2 Placebo Capsules Daily
  Other Names: Placebo
  Groups: Control - Placebo
Dietary Supplement: Group1 — Participants will receive 1 Uqora Drink-Mix and 2 Placebo Capsules Daily
  Groups: Group 1
Dietary Supplement: Group 2 — Participants will receive 1 Uqora Drink-Mix and 2 Uqora Capsules Daily
  Groups: Group 2

SUMMARY:
This is a virtual study which will invite females over the age of 18 who have had 2 or more UTIs in the past 6 months to participate. The investigators are looking at the impact of a daily dietary supplement with the recurrence of UTIs. Participants will be blinded and randomized randomized into the Control Group or Groups 1 or 2. Control Group will receive a Placebo Drink-Mix and Placebo Capsules. Group 1 will receive the Uqora Drink-Mix and Placebo Capsules. Group 2 will receive the Uqora Drink-Mix and Uqora Capsules. Each group will receive 180 day supply of the products.

DETAILED DESCRIPTION:
Urinary Track Infections (UTIs) are the second most common infection in the United Stated. There is growing concern about the amount of antibiotic use and drug resistance. Patients with frequent UTIs are encouraged to keep well hydrated. Some are encouraged to drink cranberry juice or cranberry extract. In 2016 a published study demonstrated no difference. The investigators hypothesize that the Uqora dietary supplement will decrease the frequency of UTIs.

The study was designed as a prospective randomized blinded study. Results will be patient reported results along with any confirmation of a documented UTI. Participants will be asked to keep a weekly diary logging the supplement intake. The participant will also be asked to complete the King's Health Questionnaire, a urinary health questionnaire and quality of life. The data will be entered by the participant into a portal using a personalized login and password.

ELIGIBILITY:
Inclusion Criteria:

* Is female
* Is 18 years of age or older
* Is able to swallow pills
* Has been treated with antibiotics for 2 or more UTIs in the past 6 months
* Is otherwise in good health Subjects will be deemed to be in good health if they do not report any of the existing medical conditions asked about in the screening questionnaire.

Exclusion Criteria:

* Has any of the following medical conditions: multiple sclerosis; diabetes; chronic kidney stones ○ Subjects with multiple sclerosis, diabetes, and/ or chronic kidney stones will be excluded from the study because these subjects are more likely to have complicated UTIs.
* Uses a wheelchair ○ Subjects that use a wheelchair will be excluded from the study as these subjects are more likely to have complicated UTIs.
* Regularly uses a catheter

  ○ Subjects that use catheters will be excluded from the study as these subjects are more likely to have complicated UTIs.
* Is pregnant

  ○ Pregnant women and women that become pregnant will be excluded from the study because of an increased likelihood these subjects will drop out from the study on recommendation from their physicians or other healthcare provider.
* Is currently taking Uqora brand products for UTI prevention

  ○ Subjects will be asked if they are currently taking other products for UTI prevention. If the subject indicates she is currently taking a Uqora product, she will be excluded from the study. If the subject indicates she is taking additional products for prevention (not Uqora products), she will not be excluded from the study and she will be eligible to be enrolled and randomly assigned into 1 of the 3 groups.
* Is currently taking antibiotics prophylactically for the purpose of UTI prevention ○ These subjects will be excluded from the study because they have been instructed by their physician or other healthcare provider to take antibiotics on an ongoing basis, which would have a significant impact on the recurrence of UTIs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender as diagnosed at birth without any alterations at the time of enrollment
Study Population: The study will consist of 360 female subjects aged 18 and older with at least 2 UTIs in the past 6 months. The subjects will be otherwise healthy. The geography of subject enrollment will be spread across the United States.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Recurrence of UTIs at six-months | 6-months
  A UTI is defined by the receipt of a prescription of antibiotics for treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martina Speight, MSN, FNP-BC, Principal Investigator — Hawthorne Effect Inc.
Locations (1):
- Uqora, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
The data will be owned by the Sponsor, Uqora Inc. The data will be collected, analyzed and given to the sponsor.

REFERENCES:
- [Result] Juthani-Mehta M, Van Ness PH, Bianco L, Rink A, Rubeck S, Ginter S, Argraves S, Charpentier P, Acampora D, Trentalange M, Quagliarello V, Peduzzi P. Effect of Cranberry Capsules on Bacteriuria Plus Pyuria Among Older Women in Nursing Homes: A Randomized Clinical Trial. JAMA. 2016 Nov 8;316(18):1879-1887. doi: 10.1001/jama.2016.16141. PMID 27787564
- [Result] Wullt B, Bergsten G, Samuelsson M, Svanborg C. The role of P fimbriae for Escherichia coli establishment and mucosal inflammation in the human urinary tract. Int J Antimicrob Agents. 2002 Jun;19(6):522-38. doi: 10.1016/s0924-8579(02)00103-6. No abstract available. PMID 12135844
- [Result] Bergsten G, Wullt B, Svanborg C. Escherichia coli, fimbriae, bacterial persistence and host response induction in the human urinary tract. Int J Med Microbiol. 2005 Oct;295(6-7):487-502. doi: 10.1016/j.ijmm.2005.07.008. PMID 16238023
- [Result] Altarac S, Papes D. Use of D-mannose in prophylaxis of recurrent urinary tract infections (UTIs) in women. BJU Int. 2014 Jan;113(1):9-10. doi: 10.1111/bju.12492. No abstract available. PMID 24215164
- [Result] Michaels EK, Chmiel JS, Plotkin BJ, Schaeffer AJ. Effect of D-mannose and D-glucose on Escherichia coli bacteriuria in rats. Urol Res. 1983;11(2):97-102. doi: 10.1007/BF00256954. PMID 6346629
- [Result] Ofek I, Mosek A, Sharon N. Mannose-specific adherence of Escherichia coli freshly excreted in the urine of patients with urinary tract infections, and of isolates subcultured from the infected urine. Infect Immun. 1981 Dec;34(3):708-11. doi: 10.1128/iai.34.3.708-711.1981. PMID 6120897
- [Result] Porru, D et al. "Oral D-Mannose in recurrent urinary tract infections in women - a pilot study". Journal of Clinical Urology. Volume 7, Issue 3. 2014.
- [Result] Foxman B, Chi JW. Health behavior and urinary tract infection in college-aged women. J Clin Epidemiol. 1990;43(4):329-37. doi: 10.1016/0895-4356(90)90119-a. PMID 2324774
- [Result] Ochoa-Brust GJ, Fernandez AR, Villanueva-Ruiz GJ, Velasco R, Trujillo-Hernandez B, Vasquez C. Daily intake of 100 mg ascorbic acid as urinary tract infection prophylactic agent during pregnancy. Acta Obstet Gynecol Scand. 2007;86(7):783-7. doi: 10.1080/00016340701273189. PMID 17611821
- [Result] Ebrahimi E, Khayati Motlagh S, Nemati S, Tavakoli Z. Effects of magnesium and vitamin b6 on the severity of premenstrual syndrome symptoms. J Caring Sci. 2012 Nov 22;1(4):183-9. doi: 10.5681/jcs.2012.026. eCollection 2012 Dec. PMID 25276694
- [Result] Head KA. Natural approaches to prevention and treatment of infections of the lower urinary tract. Altern Med Rev. 2008 Sep;13(3):227-44. PMID 18950249
- [Result] Yaxley, Julian. "Alkalization of urine in patients with infections of the urinary tract." British Journal of Medicine and Medical Research. 2016.
- [Result] Shields-Cutler RR, Crowley JR, Hung CS, Stapleton AE, Aldrich CC, Marschall J, Henderson JP. Human Urinary Composition Controls Antibacterial Activity of Siderocalin. J Biol Chem. 2015 Jun 26;290(26):15949-60. doi: 10.1074/jbc.M115.645812. Epub 2015 Apr 10. PMID 25861985
- [Result] Lee MJ, Maliakal P, Chen L, Meng X, Bondoc FY, Prabhu S, Lambert G, Mohr S, Yang CS. Pharmacokinetics of tea catechins after ingestion of green tea and (-)-epigallocatechin-3-gallate by humans: formation of different metabolites and individual variability. Cancer Epidemiol Biomarkers Prev. 2002 Oct;11(10 Pt 1):1025-32. PMID 12376503
- [Result] Reygaert W, Jusufi I. Green tea as an effective antimicrobial for urinary tract infections caused by Escherichia coli. Front Microbiol. 2013 Jun 18;4:162. doi: 10.3389/fmicb.2013.00162. eCollection 2013. PMID 23785367
- [Result] Packiavathy IA, Priya S, Pandian SK, Ravi AV. Inhibition of biofilm development of uropathogens by curcumin - an anti-quorum sensing agent from Curcuma longa. Food Chem. 2014 Apr 1;148:453-60. doi: 10.1016/j.foodchem.2012.08.002. Epub 2012 Aug 10. PMID 24262582
- [Result] Trujillo J, Chirino YI, Molina-Jijon E, Anderica-Romero AC, Tapia E, Pedraza-Chaverri J. Renoprotective effect of the antioxidant curcumin: Recent findings. Redox Biol. 2013 Sep 17;1(1):448-56. doi: 10.1016/j.redox.2013.09.003. PMID 24191240
- [Result] Ku, Ja Hyeon and Oh, Seung-June. Comparison of Three Quality of Life Questionnaires in Urinary Incontinence. Springer Science and Business Media. 2010.
- See also: Urinary Tract Infections — http://www.kidney.org/sites/default/files/uti.pdf
- See also: Urologic Diseases in America — http://citeseerx.ist.psu.edu/viewdoc/download?doi=10.1.1.169.5247&rep=rep1&type=pdf